CLINICAL TRIAL: NCT07069127
Title: Reduction of Dentin Hypersensitivity and Enamel Demineralization in Patients With Celiac Disease: A Randomized Controlled Trial
Brief Title: Hydroxyapatite-Based Home Treatment for Dentin Sensitivity in Celiac Patients
Acronym: CELIADENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-HApCELIAC
Record Dates: First submitted 2025-07-05; First posted 2025-07-16 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Celiac Disease; Dentin Hypersensitivity; Tooth Demineralization
Keywords: Celiac Disease; Dentin Hypersensitivity; Enamel Demineralization; Hydroxyapatite; Remineralizing Agents; Biorepair; Toothpaste; Oral Mousse; Dental Sensitivity; Randomized Controlled Trial
MeSH Terms: conditions — Celiac Disease; Dentin Sensitivity; Tooth Demineralization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biorepair Toothpaste + Mousse (Experimental): Participants in this group will perform home oral hygiene using Biorepair® Total Protection toothpaste twice daily and apply Biorepair® Plus Intensive Enamel Repair mousse once every evening before bedtime for the duration of the study (6 months).
  Interventions: Device: Biorepair Toothpaste and Mousse
- Biorepair Toothpaste Only (Active Comparator): Participants in this group will perform home oral hygiene using Biorepair® Total Protection toothpaste twice daily, without the use of the additional mousse. This regimen will continue for the entire 6-month study period.
  Interventions: Device: Biorepair® Toothpaste

INTERVENTIONS:
Device: Biorepair Toothpaste and Mousse — Participants assigned to the experimental arm will use Biorepair® Total Protection toothpaste twice daily (morning and evening) and apply Biorepair® Plus Intensive Enamel Repair mousse once daily before bedtime, for a total of 6 months. The toothpaste contains microRepair® particles (zinc-substituted hydroxyapatite), designed to occlude dentinal tubules and promote enamel remineralization. The mousse, applied at night, enhances remineralization through higher concentrations of active hydroxyapatite. This combined regimen targets the reduction of dentin hypersensitivity and enamel demineralization in adult patients with celiac disease.
  Arms: Biorepair Toothpaste + Mousse
Device: Biorepair® Toothpaste — Participants assigned to the control arm will use Biorepair® Total Protection toothpaste twice daily (morning and evening) for 6 months. The toothpaste formulation contains microRepair® (zinc hydroxyapatite) to support daily enamel protection and tubule occlusion, without the adjunctive effect of the mousse. This arm is used to assess the baseline efficacy of the toothpaste alone compared to the combined regimen.
  Arms: Biorepair Toothpaste Only

SUMMARY:
This single-center, randomized controlled clinical trial aims to evaluate the effectiveness of a home-based treatment using hydroxyapatite-based oral care products in adult patients with celiac disease who exhibit enamel demineralization and dentin hypersensitivity. Forty patients will be enrolled and randomly allocated into two parallel groups. The control group will perform home oral hygiene using only a hydroxyapatite-based toothpaste (Biorepair® Total Protection) twice daily. The trial group will follow the same regimen with the toothpaste, but will also apply a hydroxyapatite mousse (Biorepair® Plus Intensive Enamel Repair) once every evening before bedtime throughout the study period.

The primary objective is to assess the reduction in dentin hypersensitivity using the Schiff Air Index. Secondary outcomes include changes in plaque accumulation (Plaque Index), gingival bleeding (Bleeding on Probing), pain perception (Visual Analogue Scale), and caries experience (DMFT and DMFS indices). Enamel demineralization will be analyzed through near-infrared transillumination (DIAGNOcam), laser fluorescence (DIAGNOdent), and digital image analysis (ImageJ software).

All clinical parameters will be evaluated at baseline and after 1 week, 1 month, 3 months, and 6 months. The study seeks to determine whether the addition of a remineralizing mousse to daily oral care provides superior benefits in reducing sensitivity and improving enamel integrity in patients with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) with a confirmed diagnosis of celiac disease.
* Presence of enamel defects (hypomineralization or demineralization).
* Presence of active carious lesions.
* Self-reported dentin hypersensitivity.
* Willingness to comply with the study protocol and follow-up schedule.
* Written informed consent provided.

Exclusion Criteria:

* Age below 18 years.
* Absence of confirmed celiac disease.
* Poor compliance or low motivation to participate in a 6-month study.
* Ongoing treatment with products affecting enamel mineralization.
* Pregnancy or breastfeeding.
* Participation in another clinical trial within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in dentin hypersensitivity assessed by Schiff Air Index | Baseline (T0), 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4)
  The primary outcome is the variation in dentin hypersensitivity scores measured using the Schiff Air Index at baseline (T0), 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4). The Schiff Air Index is a validated clinical scale ranging from 0 to 3, where higher scores indicate greater sensitivity. The primary analysis will compare the change in scores over time between the experimental group (toothpaste + mousse) and the control group (toothpaste only).

SECONDARY OUTCOMES:
Change in plaque accumulation assessed by Plaque Index (PI) | Assessed at baseline (T0), and at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4) from the start of treatment.
  Plaque accumulation will be assessed using the Plaque Index (PI) at each time point. The index evaluates four surfaces per tooth and assigns a score from 0 to 3, where 0 indicates no plaque, 1 denotes plaque detectable only with a disclosing agent, 2 represents plaque visible to the naked eye, and 3 corresponds to abundant plaque covering the tooth surface. The average PI score per patient will be calculated and compared between the two groups over time (T0 to T4) to evaluate the impact of the interventions on daily oral hygiene and biofilm control.
Change in gingival bleeding assessed by Bleeding on Probing (BoP) | Evaluated at baseline (T0), and at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after treatment initiation.
  Gingival bleeding will be evaluated using the Bleeding on Probing (BoP) index, where gentle probing is performed and bleeding is recorded as either absent (score 0) or present (score 1). The percentage of bleeding sites per participant will be calculated, and reductions in this percentage will indicate improvements in periodontal health.
Change in self-reported pain using Visual Analogue Scale (VAS) | Measured at baseline (T0), and at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4) from the beginning of the intervention.
  Dentin hypersensitivity will be self-assessed by participants using a Visual Analogue Scale (VAS), consisting of a 10 cm line anchored at 0 (no pain) and 10 (worst imaginable pain). The score, measured in millimeters from the 0 mark, provides a quantitative measure of pain intensity. Changes in VAS scores over time will be analyzed between groups.
Change in caries experience using DMFT Index | Assessed at baseline (T0), and at follow-up visits at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4).
  The DMFT index records the total number of Decayed, Missing, and Filled permanent Teeth per individual. Scores range from 0 (no caries experience) up to 28 or 32, depending on the number of teeth present. A reduction or stabilization of DMFT scores over time will indicate an improvement or prevention of caries progression.
Change in caries experience using DMFS Index | Recorded at baseline (T0), and at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after enrollment.
  The DMFS index expands the DMFT to include all tooth surfaces, providing a more sensitive measure of caries experience. Each surface is assessed individually, and scores range from 0 (no affected surfaces) to a maximum depending on the total number of tooth surfaces. Higher values indicate more extensive caries. Scores will be compared across time points between groups.
Change in enamel lesion area assessed by DIAGNOcam and ImageJ software | Evaluated at baseline (T0), and at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4) from treatment initiation.
  The extent of enamel demineralization will be assessed using near-infrared light transillumination with the DIAGNOcam device. The captured images will be processed using ImageJ software to quantify the surface area of enamel lesions in square millimeters. Each lesion will be manually outlined and analyzed by a calibrated examiner. The score assigned will represent the total area (in mm²) of demineralized enamel per tooth. Higher values indicate greater lesion extension. A progressive reduction in lesion surface area over time will be interpreted as a sign of remineralization. Intergroup comparisons will assess the impact of the hydroxyapatite-based intervention on enamel integrity.
Change in enamel fluorescence using DIAGNOdent | Obtained at baseline (T0), and at follow-up evaluations at 1 week (T1), 1 month (T2), 3 months (T3), and 6 months (T4) following the start of treatment.
  Enamel demineralization will be measured using the DIAGNOdent pen, which emits a low-power laser and detects fluorescence from porous enamel. Each site will receive a numerical score ranging from 0 to 99, where 0-10 indicates sound enamel, 11-20 indicates initial demineralization, 21-30 suggests moderate demineralization, and scores above 30 reflect advanced mineral loss. For each lesion, the highest DIAGNOdent value will be recorded, and the average value per participant will be calculated. A reduction in fluorescence values across time points will indicate enamel remineralization and clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.